CLINICAL TRIAL: NCT03305692
Title: Optimization of New CRT Recipients: Subjects Randomized to ECG Belt or Echocardiographic Optimization
Brief Title: ECG Belt vs. Echocardiographic Optimization of CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alan J. Bank, MD (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Alan J. Bank, MD, Medical Director of Research - United Heart & Vascular Clinic, Allina Health System
Organization: Allina Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERP 3890
Record Dates: First submitted 2017-09-26; First posted 2017-10-10 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure, Systolic
Keywords: cardiac resynchronization therapy; pacing; echocardiography; optimization; heart failure
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Outcomes Assessor
Masking Description: Individual analyzing echocardiograms (primary outcome) will not know randomization of the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ECG Belt (Experimental): Use ECG Belt body surface mapping system to optimize CRT programming.
  Interventions: Diagnostic Test: Optimization of CRT Device
- Echocardiography (Experimental): Use mitral inflow echocardiography to optimize CRT programming.
  Interventions: Diagnostic Test: Optimization of CRT Device

INTERVENTIONS:
Diagnostic Test: Optimization of CRT Device — Use a body surface mapping system to quantify electrical dyssynchrony or echocardiography to quantify diastolic blood flow characteristics. Program the pacemaker to maximize the benefit of the modality the subject is randomized to.

SUMMARY:
Cardiac resynchronization therapy (CRT) has been a valuable intervention for patients with systolic heart failure for over 15 years. Despite years of research, there is a still a 25-40% non-responder rate depending on the outcomes measured. CRT optimization is a term used to describe the act of individualizing the therapy (CRT programming) for an individual patient. This is not often performed, but when it is, echocardiography is utilized. Recent work of body surface mapping using a novel system called the ECG Belt has shown a relationship between measures of electrical dyssynchrony and acute and chronic heart pumping function. This study will compare outcomes of patients randomized to either echocardiographic or ECG Belt optimization of CRT devices.

DETAILED DESCRIPTION:
This is a prospective randomized study designed to determine whether cardiac resynchronization therapy (CRT) device programming guided by the ECG Belt (Medtronic, PLC) improves echocardiographic and functional outcomes in heart failure (HF) patients. The population will include patients treated with CRT for standard indications (not implanted for the sole purposes of this study). The study will focus enrollment on patients who do not have baseline characteristics predicting the best CRT response. Therefore the study will not enroll patients having non-ischemic HF etiology, left bundle branch (LBBB) morphology, and QRSd > 150 ms or those previously RV paced.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent for participation in the study
* Age ≥18 years
* Received a first-time CRT device for standard clinical indication (can be upgraded from non-CRT pacemaker or defibrillator if ventricular pacing < 10%)
* Adequate echocardiographic images for EF & LVESV determination

Exclusion Criteria:

* Unhealed open wounds on the torso and/or a history of documented severe allergic reactions from ECG electrode gel
* Enrollment in a concurrent study that could confound the results of this study
* Pregnant or could become pregnant within the 6 month follow-up period
* Non-ischemic cardiomyopathy, LBBB morphology, and QRSd > 150 ms
* Dysrhythmia (AF or PVCs) that will likely result in aggregate ventricular pacing < 90% over the 6 month follow-up period

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Echocardiographic assessment of LV function | 6 months post optimization
  Change in ejection fraction
Echocardiographic assessment of LV size | 6 months post optimization
  Change in left ventricular end-systolic volume

CONTACTS AND LOCATIONS:
Overall Officials: Alan Bank, MD, Principal Investigator — United Heart & Vascular Clinic - Allina Health System
Locations (1):
- United Heart & Vascular Clinic, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers.